CLINICAL TRIAL: NCT06630988
Title: Diagnostic and Management of Hand Infection: a Retrospective Cohort in a Tertiary Care Center.
Brief Title: Diagnostic and Management of Hand Infection.
Acronym: HandInf
Status: Active, not recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 24-5342
Record Dates: First submitted 2024-09-26; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Hand Infections; Including Whitlows; Tendinous Infections; Septic Arthritis
Keywords: Hand infection; Whitlows; Tendinous infections; Septic arthritis
MeSH Terms: conditions — Arthritis, Infectious

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Hand infection: Description of whitlows, tendinous infections and septic arthritis diagnostic, management and outcome Descriptive study, no intervention
  Interventions: Other: Failure rates

INTERVENTIONS:
Other: Failure rates — Describe the management failure rate for hand infections, including panariasis, phlegmons and arthritis.

SUMMARY:
Primary or secondary (post-traumatic infections, notably related to bites, wounds, etc.) infections of the hand are very common situations, even if the epidemiology is poorly understood. For example, hand bite injuries represent 1.2 million referrals to the healthcare system per year in the United States. Their nosological framework extends from simple infections of the skin and soft tissues such as whitlows, to potentially severe deep damage such as arthritis and osteitis, or phlegmons of the tendon sheaths. The diagnostic approach is not consensual, and the contribution of additional biological parameters (inflammatory syndrome) and morphological investigations (x-rays, ultrasound, CT-scan or MRI) is not codified. Microbiology seems dominated by Staphylococcus aureus, but few studies have precisely described the microbial etiology. Consequently, probabilistic antibiotic therapy and the need to take bacteriological samples for secondary adaptation are not standardized. Likewise, surgical strategies (abstention, systematic washing or depending on evolution) remain operator dependent. We consequently aim to described diagnostic, management and related outcomes or hand infections in a specialized tertiary care center.

ELIGIBILITY:
Inclusion Criteria:

* all patient ≥ 18
* yo followed-up for a hand infection in our tertiary care center
* from 01/01/2014 to 31/12/2023, including
* whitlows
* tendinous infections
* septic arthritis

Exclusion Criteria:

* osteomyelitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be selected from the data base of the hand emergency surgery department of our tertiary care center, based on a principal or secondary diagnosis of BJI appearing alone or in combination with either sepsis or a specific surgical procedure - 1400 potential patients.
Sampling Method: Non-Probability Sample
Enrollment: 1400 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of treatment failure during the management of hand infections. | between 01/01/2014 and 31/12/2023.
  Treatment failure will be defined as infection persistence or relapse, need of unplanned surgery for septic reason or infection-related death.

CONTACTS AND LOCATIONS:
Overall Officials: Florent Valour Pr Florent Valour, Pr, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- HCL - Hôpital Edouard Herriot, Lyon, France